CLINICAL TRIAL: NCT00830999
Title: VLDL-triglyceride Metabolism in Response to Acute Diet- and Exercise-induced Changes in Energy Balance
Brief Title: Fat Metabolism in Response to Acute Diet- and Exercise-induced Changes in Energy Balance
Acronym: DEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0195
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases
Keywords: fat metabolism; exercise; liver; lipoproteins; triglycerides
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Positive energy balance (Experimental): Comparison between isocaloric and hypercaloric diets with no exercise performed in any trials
  Interventions: Behavioral: Positive energy balance; Behavioral: Energy balance
- Energy balance with exercise (Experimental): Comparison between an isocaloric diet without exercise and a hypercaloric diet with a sufficient amount of exercise performed to match the excess calories consumed resulting in both trials being in net energy balance.
  Interventions: Behavioral: Energy balance with exercise; Behavioral: Energy balance
- Negative energy balance (Experimental): Comparison between isocaloric and hypocaloric diets with no exercise performed in any trials
  Interventions: Behavioral: Negative energy balance; Behavioral: Energy balance
- Negative energy balance with exercise (Experimental): Comparison between consuming an isocaloric diet without exercise and consuming the same amount of calories as in the isocaloric trial but with exercise performed resulting in net negative energy balance in the exercise trial.
  Interventions: Behavioral: Negative energy balance with exercise; Behavioral: Energy balance

INTERVENTIONS:
Behavioral: Positive energy balance — Subjects will consume over a 24 hour period 33% more calories than they require to meet their energy demands.
  Arms: Positive energy balance
Behavioral: Energy balance with exercise — Subjects will consume over a 24 hour period 33% more calories than they require to meet their energy demands but will perform 2 hours of exercise that will be sufficient to burn off the excess calories consumed resulting in subjects being in net energy balance.
  Arms: Energy balance with exercise
Behavioral: Negative energy balance — Subjects will consume over a 24 h period only 66% of the calories required to meet their energy demands such that they will be in a net negative calorie balance in this trial.
  Arms: Negative energy balance
Behavioral: Negative energy balance with exercise — Subjects will consume over a 24 hour period the same amount of calories as ingested in the isocaloric trial but will also perform 2 hours of exercise that will be sufficient to burn off a third of the calories they consumed during this day resulting in subjects being in net negative energy balance in this trial
  Arms: Negative energy balance with exercise
Behavioral: Energy balance — Subjects will consume over a 24 hour period a sufficient amount of calories to meet their energy needs.

SUMMARY:
This study is being conducted to learn more about the role of diet and exercise in regulating plasma triglyceride (fat) metabolism. The investigators will examine the effect of acute (24 hour) changes in energy intake and expenditure on fat metabolism the following day.

DETAILED DESCRIPTION:
Excess body fat and a sedentary lifestyle are associated with increased plasma triglyceride (TG) and apolipoprotein B-100 (apoB-100) concentrations, which are important risk factors for the development of cardiovascular disease.

Weight loss and endurance exercise improve plasma lipid and lipoprotein concentrations. However, the mechanisms responsible for this effect are largely unknown, and much uncertainty remains regarding the independent roles of dietary energy intake, exercise energy expenditure, and net energy balance in controlling plasma TG concentrations.

The main goal of this project, therefore, is to investigate the mechanisms by which acute alterations in energy balance, induced by diet and/or physical activity (endurance exercise), regulate very-low density lipoprotein (VLDL) metabolism.

Subjects will be asked to perform 3 separate trials. One of these will always be an "energy balance" trial that will act as the control trial for the other 2 trials they perform. Subjects will therefore be randomized to 2 different study arms.

ELIGIBILITY:
Inclusion Criteria:

* overweight and obese men
* normal to mild hypertriglyceridemia

Exclusion Criteria:

* Smoking
* Any medical condition other than increased body weight (e.g. diabetes, heart disease, etc.).
* Use of drugs known to affect lipid metabolism (e.g. statins, etc.).
* Regular exercise training.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Very Low Density Lipoprotein-Triglyceride and apoB-100 concentrations | After acute (24 hour) changes in energy intake and/or energy expenditure

SECONDARY OUTCOMES:
Liver Very Low Density Lipoprotein-Triglyceride and apoB-100 secretion rates | After acute (24 hour) changes in energy intake and/or energy expenditure
Liver Very Low Density Lipoprotein-Triglyceride and apoB-100 clearance rates from plasma | After acute (24 hour) changes in energy intake and/or energy expenditure
Plasma glucose concentration and turnover rate | After acute (24 hour) changes in energy intake and/or energy expenditure
Plasma insulin concentration | After acute (24 hour) changes in energy intake and/or energy expenditure
Plasma free fatty acid concentration and turnover rate | After acute (24 hour) changes in energy intake and/or energy expenditure
Plasma glucose concentration | During acute (24 hour) changes in energy intake and/or energy expenditure
  Measured hourly over the 24 h period.
Plasma insulin concentration | During acute (24 hour) changes in energy intake and/or energy expenditure
  Measured hourly over the 24 h period.
Plasma free fatty acid concentration | During acute (24 hour) changes in energy intake and/or energy expenditure
  Measured hourly over the 24 h period.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

REFERENCES:
- [Derived] Smith GI, Magkos F, Reeds DN, Okunade AL, Patterson BW, Mittendorfer B. One day of mixed meal overfeeding reduces hepatic insulin sensitivity and increases VLDL particle but not VLDL-triglyceride secretion in overweight and obese men. J Clin Endocrinol Metab. 2013 Aug;98(8):3454-62. doi: 10.1210/jc.2013-1786. Epub 2013 Jun 7. PMID 23750033